CLINICAL TRIAL: NCT02372929
Title: Relationship Between Endoscopic Ultrasound Staging and Degree of Stricture in Esophageal Cancer
Acronym: ESOCA
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 356407
Record Dates: First submitted 2015-02-16; First posted 2015-02-26 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2017-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic Ultrasound Staging: Prospective study of esophageal cancer patients referred for endoscopic ultrasound
  Interventions: Procedure: Endoscopic Ultrasound

INTERVENTIONS:
Procedure: Endoscopic Ultrasound — Esophageal cancer patients will be staged by endoscopic ultrasound. All patients will undergo upper endoscopy prior to endoscopic ultrasound.

SUMMARY:
The primary objective of this study is to document all cases of EUS in patients with esophageal cancer and determine if the inability to advance the gastroscope beyond the tumor correlates with locally advanced disease stage at Endoscopic Ultrasound.

DETAILED DESCRIPTION:
This will be an observational prospective study. The investigators will aim to enroll 100 male and female adult patients (aged 19 years and over) of all ethnicities/races, who have been referred to Florida Hospital for Endoscopic Ultrasound staging of esophageal cancer. All vulnerable populations will be excluded.

The investigators will be using a standardized data collection form to record presenting symptoms, endoscopy findings, Endoscopic Ultrasound features and final esophageal cancer staging. This is an observational study in which standard of care is being practiced and also as the patients are not placed at additional risk from participating in this study. However, as the investigators are collecting data prospectively, all participants will sign consent. An attempt will be made to see if there is a correlation between stricture tightness encountered at endoscopy (EGD) with advanced disease stage diagnosed at Endoscopic Ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1.All patients aged > 18 yrs, who can provide informed consent and referred to Florida Hospitals Endoscopy Unit for EUS staging of esophageal cancer.

Exclusion Criteria:

1. Age < 18 yrs
2. Inability to provide informed consent.
3. Unable to safely undergo endoscopy for any reason
4. Coagulopathy (prolongation of Prothrombin time > 18 secs, thrombocytopenia < 80,000 platelets/ml)
5. Limited mental capacity or language skills to the extent simple instructions cannot be followed or information regarding adverse events and follow-up phone visits cannot be provided
6. Non-English speaking without a translator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for EUS for esophageal cancer staging will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the relationship between tightness of esophageal stricture encountered at endoscopy with cancer staging at EUS. | Intraoperative
  The investigators hypothesize that if the stricture (cancer) in the esophagus is high-grade it will preclude passage of the endoscope and subjects on endoscopic ultrasound are likely to have advance-stage disease. An attempt will be made to correlate the relationship between stricture tightness and disease stage of esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam S Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital Center for Interventional ENdoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript will be developed upon completion of the study